CLINICAL TRIAL: NCT00662311
Title: Phase I/II Clinical Trial Evaluating the Use of Vorinostat Combined With Paclitaxel and Radiotherapy in Patients With Inoperable Stage III Non-Small Cell Lung Cancer Unable to Tolerate Cisplatin
Brief Title: Vorinostat, Paclitaxel, and Radiation Therapy in Treating Patients Unable to Tolerate Cisplatin With Stage III Non-Small Lung Cancer That Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shilpen Patel, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6600; NCI-2010-00715 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Paclitaxel; Taxes; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (vorinostat with paclitaxel and radiotherapy) (Experimental): Patients receive vorinostat PO QD, 5 days a week and paclitaxel IV over 1 hour once a week. Patients also undergo radiation therapy QD, 5 days a week. Treatment repeats every week for 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
This phase I/II trial studies the side effects and best dose of vorinostat when given together with paclitaxel and radiation therapy and to see how well it works in treating patients unable to tolerate cisplatin with stage III non-small cell lung cancer (NSCLC) that cannot be removed by surgery. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving vorinostat together with paclitaxel and radiation therapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of vorinostat when administered in combination with paclitaxel and thoracic radiation therapy in patients with locally advanced NSCLC.

SECONDARY OBJECTIVES:

I. To assess the safety and toxicity of vorinostat when administered in combination with paclitaxel and thoracic radiation therapy in patients with locally advanced NSCLC.

II. To determine the radiological response rate, by computed tomography (CT) scan, of vorinostat when administered in combination with paclitaxel and thoracic radiation therapy in patients with locally advanced NSCLC.

III. To describe the progression free survival (PFS) and overall survival (OS) of this regiment over 3 years of follow up.

OUTLINE: This is a phase I, dose-escalation study of vorinostat followed by a phase II study.

Patients receive vorinostat orally (PO) once daily (QD), 5 days a week and paclitaxel intravenously (IV) over 1 hour once a week. Patients also undergo radiation therapy QD, 5 days a week. Treatment repeats every week for 7 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 12 weeks, every 3 months for 2 years, and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of NSCLC
* Inoperable Stage IIIA or IIIB (excluding malignant pleural effusion) disease according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual, Sixth edition (2002)
* At least one site of measurable disease, as defined by the modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Inability to tolerate full dose cisplatin as defined by:
* Creatinine clearance less than 50ml/min
* Greater than grade 2 sensory hearing loss (as defined by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] criteria v3.0 adverse event term "Hearing: Patients without baseline audiogram and not enrolled in a monitoring program")
* Performance status >= 2
* Age >= 75 years
* Cardiac history, such as myocardial infarction within 6 months, angina, or heart disease as defined by the New York Heart Association (NYHA) Class III or IV
* Any other comorbid disease or condition that would increase the risk of toxicity of cisplatin therapy
* Female patient is either post menopausal, free from menses for >= 2 years, surgically sterilized or willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual activity throughout the study
* Female patient of childbearing potential has a negative serum pregnancy test beta-human chorionic gonadotropin (hCG) within 7 days prior to receiving the first dose of vorinostat
* Male patient agrees to use an adequate method of contraception for the duration of the study
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Prothrombin Time or International Normalized Ratio (INR) =< 1.5x upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) =< 1.2 times the ULN unless the patient is receiving therapeutic anticoagulation
* Potassium levels: Normal limits
* Magnesium levels: Normal limits
* Calculated creatinine clearance >= 20 mL/min
* Serum total bilirubin =< 1.5 X ULN
* Aspartate aminotransferase (AST) (serum glutamate oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN
* Alkaline Phosphatase =< 2.5 X ULN
* Patient, or the patient's legal representative, has voluntarily agreed to participate by giving written informed consent
* Patient has a life expectancy of at least 12 weeks
* Patient is available for periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study

Exclusion Criteria:

* Patient who has had chemotherapy, radiotherapy, or biological therapy for NSCLC within 5 years prior to initial dosing with study drug(s)
* Symptomatic neuropathy (>= grade 2)
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drug(s)
* Patient had prior treatment with an histone deacetylases (HDAC) inhibitor (e.g., romidespsin [Depsipeptide, NSC-630176], entinostat [MS 275], dacinostat [LAQ-824], belinostat [(PXD-101]), panobinostat [LBH589], mocetinostat [MGCD0103], CRA024781, etc); patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study; patients who have received such compounds for other indications, e.g., valproic acid for epilepsy, may enroll after a 30-day washout period
* Patient has known hypersensitivity to the components of study drug or its analogs or paclitaxel
* NYHA Class III or IV congestive heart failure, myocardial infarction within the previous 6 months, QTc > 0.47 seconds, or uncontrolled arrhythmia
* Patient is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study
* Patient with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled; patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for > 5 years or are considered by their physician to be at less than 30% risk of relapse
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shilpen Patel, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat 200 mg: Cohort 1: Patients receive 200 mg vorinostat PO QD, 5 days a week and paclitaxel IV over 1 hour once a week. Patients also undergo radiation therapy QD, 5 days a week. Treatment repeats every week for 7 courses in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given PO
  paclitaxel: Given IV
  radiation therapy: Undergo radiation therapy
- Vorinostat 300 mg: Cohort 2: Patients receive 300 mg vorinostat PO QD, 5 days a week and paclitaxel IV over 1 hour once a week. Patients also undergo radiation therapy QD, 5 days a week. Treatment repeats every week for 7 courses in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given PO
  paclitaxel: Given IV
  radiation therapy: Undergo radiation therapy
- Vorinostat 400 mg: Cohort 3: Patients receive 400 mg vorinostat PO QD, 5 days a week and paclitaxel IV over 1 hour once a week. Patients also undergo radiation therapy QD, 5 days a week. Treatment repeats every week for 7 courses in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given PO
  paclitaxel: Given IV
  radiation therapy: Undergo radiation therapy
Period: Overall Study
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg
Started | 5 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Respiratory Infection | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat 400 mg: Cohort 3: Patients receive 300 mg vorinostat PO QD, 5 days a week and paclitaxel IV over 1 hour once a week. Patients also undergo radiation therapy QD, 5 days a week. Treatment repeats every week for 7 courses in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given PO
  paclitaxel: Given IV
  radiation therapy: Undergo radiation therapy
- Total: Total of all reporting groups
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg | Total
Number analyzed (Participants) | 5 | 0 | 0 | 5
Age, Continuous [Mean (Full Range); unit: years] | 77 [74 to 80] |  |  | 77 [74 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  | 3
  Male | 2 |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 5 |  |  | 5
  Unknown or Not Reported | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: MTD of Vorinostat When Administered in Combination With Paclitaxel and Radiotherapy Therapy as Assessed by NCI Common Toxicity Criteria for Adverse Events (CTCAE) Version 3.0 (Phase I)
Description: Defined as the highest dose level at which no more than 1 of 6 patients experiences dose-limiting toxicity (DLT). Toxicity was graded according to the National Institutes of Health Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. A DLT was defined as any Grade 3 or higher non-hematologic adverse event with the exception of alopecia, fatigue, or anorexia. Nausea and/or vomiting that persisted > 48 hours despite optimal medical management at grade 3 or higher was considered a DLT. Hematologic dose-limiting toxicity was defined as either: Grade 4 neutropenia lasting for ≥ 7 days in duration, Grade > 3 febrile neutropenia with/without infection, Grade 4 thrombocytopenia or Grade 5 hematologic toxicity.
Time Frame: 8 weeks
Measure: Number; unit: mg
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg
Number analyzed (Participants) | 5 | 0 | 0
mg | NA — Due to adverse events we were unable to increase the vorinostat dosing beyond the first cohort of 200mg. The study was terminated prior to identifying the MTD. |  |

2. Secondary Outcome: Radiological Response Rate as Assessed by CT
Description: Count of participants with stable disease or partial response. Patients were evaluated for treatment response per RECIST criteria (version 1.0).
Time Frame: 12 weeks post-treatment, then every 3 months for 2 years, and then every 6 months for a year thereafter
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg
Number analyzed (Participants) | 5 | 0 | 0
Participants
  12 Weeks | 4 |  |
  6 Months | 3 |  |
  9 Months | 3 |  |
  12 Months | 1 |  |
  15 Months | 1 |  |
  18 Months | 1 |  |
  21 Months | 1 |  |
  24 Months | 1 |  |
  27 Months | 1 |  |
  33 Months | 0 |  |
  39 Months | 0 |  |

3. Secondary Outcome: Duration of Response
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg
Number analyzed (Participants) | 4 | 0 | 0
months | 10 [6 to 28.2] |  |

4. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier estimate. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0).
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: progression free survival probability
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg
Number analyzed (Participants) | 5 | 0 | 0
progression free survival probability | 0.20 [0.035 to 1.00] |  |

5. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimate
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg
Number analyzed (Participants) | 5 | 0 | 0
survival probability | 0.60 [0.29 to 1.00] |  |

6. Secondary Outcome: Safety and Toxicity of Vorinostat at the MTD as Assessed by NCI CTCAE Version 3.0
Description: Count of participants with a grade 3 or higher toxicity. Toxicities were assessed using the NCI CTCAE (v3.0). Grade 3 or higher toxicities were considered worse.
Time Frame: Weekly during treatment, 30 days post-treatment, and 12 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg
Number analyzed (Participants) | 5 | 0 | 0
Participants | 4 |  |

ADVERSE EVENTS:
Arm/Group | Vorinostat 200 mg | Vorinostat 300 mg | Vorinostat 400 mg
Serious Adverse Events (participants affected / at risk) | 4/5 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat 200 mg (N=5) | Vorinostat 300 mg (N=0) | Vorinostat 400 mg (N=0)
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Community Contacted Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Radiation Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes